CLINICAL TRIAL: NCT07371767
Title: A Prospective, Single-center, Open-label, Single-arm Clinical Study to Evaluate the Safety and Efficacy of CS-121, an In Vivo Base Editing Therapy Delivered by Lipid Nanoparticles Targeting APOC3, in Children and Adolescents With Hyperchylomicronemia
Brief Title: CS-121 APOC3 Base Editing in Children and Adolescents With Hyperchylomicronemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: CorrectSequence Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, Xiumin Wang, PhD, chief physician, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS-121-02
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hyperchylomicronemia
Keywords: Acute Pancreatitis; Apolipoprotein C3 (APOC3); In Vivo Base Editing; Lipid Nanoparticles (LNP); Gene Editing Therapy; Children and Adolescents
MeSH Terms: conditions — Hyperlipoproteinemia Type I; Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low Dose CS-121 (Experimental): Participants in this arm will receive low dose of CS-121
  Interventions: Biological: CS-121
- Middle Dose CS-121 (Experimental): Participants in this arm will receive middle dose of CS-121
  Interventions: Biological: CS-121
- High Dose CS-121 (Experimental): Participants in this arm will receive high dose of CS-121
  Interventions: Biological: CS-121

INTERVENTIONS:
Biological: CS-121 — CS-121 is a in vivo base editing therapy formulated in lipid nanoparticles for targeted editing of the APOC3 gene in hepatocytes.

SUMMARY:
This is a Prospective, Single-center, Open-label, Single-arm Clinical Study to Evaluate the Safety and Efficacy of CS-121, an In Vivo Base Editing Therapy Delivered by Lipid Nanoparticles Targeting APOC3, in Children and Adolescents (4-18 years) With Hyperchylomicronemia

DETAILED DESCRIPTION:
CS-121 is an investigational, in vivo base editing therapy delivered by lipid nanoparticles (LNPs) targeting the APOC3 gene in the liver. By introducing precise base edits at specific APOC3 loci, CS-121 is intended to mimic naturally occurring protective mutations that reduce APOC3 expression, thereby restoring triglyceride clearance pathways and lowering pancreatitis risk. Preclinical studies in transgenic mouse and non-human primate models demonstrated dose-dependent APOC3 editing, reductions in serum ApoC3 protein and triglyceride levels, and acceptable safety profiles, supporting advancement into human evaluation. This open-label, single-arm, dose-escalation early exploratory trial designed to evaluate the safety, tolerability, PK/PD characteristics and preliminary efficacy of CS-121 in patients with hyperchylomicronemia. Based on the properties of gene editing therapy, the primary focus of the study is to identify the optimal biological dose (OBD) rather than the traditional maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 4 years ≤ age < 18 years.
* Severe hypertriglyceridemia (sHTG), defined as a triglyceride (TG) level ≥ 500 mg/dL.
* Confirmed diagnosis of genetically inherited FCS via genetic testing, or clinically diagnosed FCS plus persistent chylomicronemia.
* Failure to achieve adequate TG control, For participants under 8 years of age, the investigator determine at their discretion whether prior lipidlowering therapy has been administered.
* Participants aged 6 years and above must sign the informed consent form themselves; for participants under 18 years of age, their parent/legal guardian must sign the informed consent form. (Participants under 6 years of age are exempt from signing the written informed consent form).
* Female participants of childbearing potential must have a negative result on serum pregnancy testing.

Exclusion Criteria:

* Currently participating in other interventional clinical studies, or having an insufficient washout period of less than 5 half-lives or 30 days (whichever is longer) since the last administration of other investigational drugs.
* Used antisense oligonucleotide (ASO)-based or small interfering RNA (siRNA)-based lipid-lowering drugs targeting APOC3 within 3 months prior to study drug administration.
* History of acute pancreatitis within 1 month before dosing.
* Patients who underwent major surgery within 3 months prior to study drug administration and are judged by the investigator as unsuitable for receiving the study drug, due to potential intolerance to adverse events such as cytokine release storm.
* ALT or AST ≥2 × ULN
* Total bilirubin ≥1.5 × ULN
* eGFR <30 mL/min/1.73 m²
* Random urine albumin-to-creatinine ratio (UACR) >30 mg/g, or urine protein is ≥ 2+
* HbA1c ≥9%
* Coagulation function abnormalities judged by the investigator as unsuitable for CS-121 administration.
* Positive results for HBsAg, dual positivity for HCV antibody and RNA, positive for HIV, or positive for Treponema pallidum infection.
* Known major organ diseases, mental disorders, Cushing's syndrome, hypothyroidism, history of lymphoproliferative disorders, or malignant tumors in any organ system, which are judged by the investigator as unsuitable for study participation due to potential intolerance to adverse events such as cytokine Release-Storm.
* Concomitant medications/treatments judged by the investigator to affect lipid metabolism, liver and kidney function, coagulation function, or interfere with the efficacy evaluation of the study drug.
* Patients of childbearing potential who are planning pregnancy, breastfeeding, or have fertility plans.
* History of hypersensitivity to any study drug, its excipients, or drugs of similar chemical classes.
* Other medical conditions or comorbidities that, in the investigator's opinion, may interfere with study compliance or data interpretation.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2041-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | Within 14 days post CS-121 dosing
The incidence and severity of treatment-emergent adverse events (TEAEs) | from screening to 10 months post last dosing

SECONDARY OUTCOMES:
Changes in serum triglyceride (TG) levels | From baseline to 10 months post last dosing
Changes in serum ApoC3 levels from baseline | From baseline to 10 months post last dosing
Concentrations of the active components of CS-121 (sgRNA and mRNA) | From baseline to 1 month post last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Children's Medical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided